CLINICAL TRIAL: NCT03132285
Title: Safety and Acceptability Study of Non-Surgical Male Circumcision Device for Adult Male Population When Removing the Foreskin Shortly After Placement of Device Performed at Lusaka and Livingstone, Zambia
Brief Title: Safety and Acceptability Study of PrePex Device When Removing the Foreskin Shortly After Placement of Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Zambia (Other Government)
Responsible Party: Principal Investigator, David Linyama, General surgeon, Ministry of Health, Zambia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2017-04-04; First posted 2017-04-27 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrePex Day 0 foreskin removal (Other): Day 0 foreskin removal
  Interventions: Device: PrePex

INTERVENTIONS:
Device: PrePex — Prepex is a non surgical male circumcision device

SUMMARY:
To assess the safety and acceptability of the non-surgical PrePex device among healthy adult male participants scheduled for voluntary medical male circumcision when removing the foreskin shortly after device placement.

DETAILED DESCRIPTION:
To assess the safety and acceptability of the non-surgical PrePex device among healthy adult male participants scheduled for voluntary medical male circumcision when removing the foreskin shortly after device placement.

Five hundred (500) males scheduled for voluntary circumcision performed by clinicians or nurses using the PrePex.

Theses clinicians and nurses have already been trained in the Prepex procedure and will undergo further training in the modification to the technique. Study duration per participant will be up to 8 weeks and will include three follow up visits and one phone call follow up.

ELIGIBILITY:
Inclusion Criteria:

* Ages - 13 to 49 years
* Uncircumcised
* Participant wants to be circumcised
* Participant assent to the procedure
* Legal guardian consent to the procedure for ages 13-18 years
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse for 8 weeks after circumcision
* Agrees to abstain from masturbation for at least 2 weeks after Removal
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 7 weeks post removal (8 weeks total)
* Participant able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study

Exclusion Criteria:

* Legal guardian withholds consent for ages 13-18 years
* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the participant from undergoing a circumcision
* Participant with the following diseases/conditions: phimosis, paraphimosis, adhesions, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Participant that to the opinion of the investigator is not a good candidate
* Diabetes Mellitus
* HIV Sero-positive

Ages: 13 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Uncircumcised males
Enrollment: 500 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2017-06-17 (Actual)

PRIMARY OUTCOMES:
Number of incidents related to the change in procedure | 8 weeks
  To assess the safety of PrePex device when removing the foreskin shortly after device placement by means of the following parameter: Incidence of Serious Adverse Events, when performed by clinicians and nurses
Acceptability of the changes procedure to patients | 8 weeks
  To asses the new procedure acceptability for patients using the following measures - Evaluation of pain during foreskin removal
  * Patients willingness to wait for foreskin removal
  * Odour while device is in situ
  * Pain at key time points on Removal visit
  * Discomfort of any type to patients.

SECONDARY OUTCOMES:
Effect of the change in procedure on circumcision healing time | 8 weeks
  To assess the circumcision healing time period.

CONTACTS AND LOCATIONS:
Locations (2):
- Zambia (2):
  - Matero Main Clinic, Lusaka, Lusaka Province
  - Dambwa North Clinic, Livingstone

IPD SHARING:
Plan to Share IPD: No